CLINICAL TRIAL: NCT01620229
Title: Maintenance Therapy With Brentuximab Vedotin (SGN-35) After Allogeneic Hematopoietic Cell Transplantation for Hodgkin Lymphoma and CD30+ Hematologic Malignancies
Brief Title: Brentuximab Vedotin After Donor Stem Cell Transplant in Treating Patients With Hematologic Malignancies
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Seagen Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2560.00; NCI-2012-00924 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2560.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); P01CA018029 (NIH)
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Hematopoietic/Lymphoid Cancer
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (brentuximab vedotin) (Experimental): Patients receive brentuximab vedotin IV on day 1. Treatment repeats every 21 days for up to 16 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: brentuximab vedotin; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: brentuximab vedotin — Given IV
  Other Names: Adcetris; anti-CD30 ADC SGN-35; anti-CD30 antibody-drug conjugate SGN-35; antibody-drug conjugate SGN-35; SGN-35
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I/II trial studies the side effects and best way to give brentuximab vedotin and to see how well it works after donor stem cell transplant in treating patients with hematologic malignancies. Monoclonal antibodies, such as brentuximab vedotin, can block cancer growth in different ways. Some block the ability of cancer to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Monoclonal antibodies may kill cancer cells that are left after donor stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the incidence of durable donor hematopoietic engraftment (defined by donor T-cell chimerism > 50% at day +84 after hematopoietic cell transplantation [HCT]) after allogeneic HCT and post-transplant brentuximab vedotin.

SECONDARY OBJECTIVES:

I. Rates of complete and partial response; incidence of acute graft-versus-host disease (GVHD) grades II-IV and chronic GVHD; overall and progression-free survival; rates of serious adverse events associated with brentuximab vedotin.

OUTLINE:

Patients receive brentuximab vedotin intravenously (IV) on day 1. Treatment repeats every 21 days for up to 16 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a cluster of differentiation (CD)30+ malignancy, with CD30 positivity demonstrated either at time of original diagnosis or at any subsequent time point
* Patients must have undergone allogeneic HCT from a related or unrelated donor; acceptable donors include:

  * Related donors: genotypically or phenotypically identical by serological typing for human leukocyte antigen (HLA)-A, -B, -C, and at the allele level for -DRB1 and -DQB1
  * Unrelated donors: Fred Hutchinson Cancer Research Center (FHCRC) matching allowed will be grade 1.0 to 2.1: matched for HLA-A, -B, -C, -DRB1 and -DQB1 by high-resolution typing
  * For all donors, a single allele disparity will be allowed for HLA-A, -B, or -C as defined by high-resolution typing
  * Patients with HLA-haploidentical donors are not eligible
* Patients must have documented post-transplant donor CD3+ chimerism of > 50% in sorted peripheral-blood CD3+ cells
* Patients must be at least 28 days out from allogeneic HCT at the time of enrollment; in general, patients should be no more than 60 days out from allogeneic HCT at time of enrollment; however, patients more than 60 days out from allogeneic HCT may be considered for enrollment in discussion with the protocol investigator (Dr. Maloney)
* Patients must be enrolled on an FHCRC non-myeloablative allogeneic transplant protocol (not standard treatment plan); for eligibility purposes, "non-myeloablative" is defined here as conditioning therapy consisting of =< 4 Gy total body irradiation, with or without fludarabine
* Patients with prior exposure to brentuximab vedotin are eligible for enrollment on this trial, regardless of previous disease response
* Women of childbearing age and men with female partners of childbearing age must be willing and able to use an effective method of contraception during the study and for at least 30 days after the last study dose of brentuximab vedotin
* Patients must be able to give informed consent

Exclusion Criteria:

* Patients who are seropositive for human immunodeficiency virus (HIV)
* Women who are pregnant or breast-feeding
* Patients with moderate to severe peripheral neuropathy (grade 2 or higher); patients with a history of moderate/severe peripheral neuropathy may be enrolled if their neuropathy improves to =< grade 1 at the time of enrollment
* Patients with significant hepatic dysfunction, as manifested by a total serum bilirubin > 4.0 g/dL; or clinical evidence of decompensated hepatic failure; or clinical evidence of decompensated portal hypertension
* Patients with an absolute neutrophil count of < 1,000 cells/mm^3
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status of > 2
* Patients with a serum creatinine > 3.0 mg/dL
* Patients with known hypersensitivity to brentuximab vedotin or any excipient contained in the drug formulation
* Patients currently receiving treatment with other systemic anti-neoplastic or investigational agents targeting their CD30+ hematologic malignancy
* Patients with active and uncontrolled infection not responding to appropriate treatment should be discussed with the study investigator (Dr. Maloney) before enrollment
* Patients who have received donor lymphocyte infusion for low donor chimerism or pending graft rejection are not eligible

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Incidence of durable hematopoietic engraftment defined as the achievement of > 50% donor CD3+ cell chimerism | At day 84 after HCT
  Evaluated according to the allogeneic transplant protocol on which patients are co-enrolled, or according to institutional standard practice if no monitoring scheme is specified in the transplant protocol.

SECONDARY OUTCOMES:
Rates of relapse | Up to 5 years
  Response criteria will be based on the 2007 revisions to the International Working Group criteria for malignant lymphoma.
Non-relapse mortality | Up to 5 years
  Response criteria will be based on the 2007 revisions to the International Working Group criteria for malignant lymphoma.
Incidence of acute GVHD | Up to 5 years
Peak grade of acute GVHD | Up to 5 years
Incidence of chronic GVHD | Up to 5 years
Severity of chronic GVHD | Up to 5 years
Incidence of adverse events related to brentuximab vedotin, graded according to National Cancer Institute Common Toxicity Criteria version 4 | Up to 30 days after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: David Maloney, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States